CLINICAL TRIAL: NCT02274870
Title: Liposomal Bupivacaine for Total Knee Arthroplasty Postoperative Analgesia
Brief Title: Liposomal Bupivacaine for Post Operative Pain After Knee Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Joseph Marino M.D., Physician, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB: 14-237B
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposome Bupivacaine, (Experimental): Liposome Bupivacaine 266mg, Knee Infiltration
  Interventions: Drug: Liposome Bupivacaine
- Bupivacaine HCl (Active Comparator): Bupivacaine HCl Continuous Femoral Nerve Block (CFNB), bolus and continuous for 48 hrs)
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Liposome Bupivacaine — Administered via local tissue infiltration around the knee joint
  Other Names: Bupivacaine Liposome, Injectable Suspension
  Arms: Liposome Bupivacaine,
Drug: Bupivacaine HCl — Administered via CFNB
  Other Names: Standard of Care
  Arms: Bupivacaine HCl

SUMMARY:
Continuous femoral nerve blocks (CFNB) provide effective pain control to patients undergoing total knee replacement (TKR). However the resulting motor blockade can lead to decreased quadriceps muscle strength and delayed functional recovery.The purpose of this study is to compare the effect of Liposome Bupivacaine infiltration into the knee to CFNB on pain control and functional recovery

DETAILED DESCRIPTION:
This is a prospective, randomized, active controlled study in patients undergoing total knee replacement. The objective of this study is to compare the efficacy of Liposome Bupivacaine, in managing postoperative pain, to standard of care CFNB. Following informed consent, patients will be randomized to one of two groups, Liposome Bupivacaine or active control, CFNB group.

266 mg Liposome Bupivacaine plus Bupivicaine HCL (150mg) will be administered via local joint infiltration around the knee joint prior to wound closure. In the control group a CFNB will be placed for 48hrs prior to surgery. Outcomes measured included pain at rest, movement and quadriceps muscle strength on the first and second postoperative day.

It is hypothesized that Liposome Bupivacaine will provide effective pain control and improved preservation of quadriceps muscle strength, in comparison to CFNB.

ELIGIBILITY:
Inclusion Criteria:

* ASA Status I-III
* Scheduled to undergo primary unilateral total knee arthroplasty

Exclusion Criteria:

* Patients who are pregnant or nursing
* Alcohol or narcotic dependence within the last 2 years
* Condition requiring regular use of analgesia that may confound post surgical assessments as determined by principle investigator
* BMI > 40kg/m2
* Contraindication to acetaminophen, morphine, oxycodone, ketorolac, epinephrine, or pathological conditions potentially aggravated by epinephrine
* Allergies to amide-type local anesthetics
* Any disease condition or lab result that could complicate a patients postoperative recovery
* History of hypotension
* Abnormal liver, renal or cardiac function
* Other physical, mental or medical conditions that, in the opinion of the investigator, make study participation inadvisable.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Marino, MD, Principal Investigator — Northwell Health
Locations (1):
- Franklin, Valley Stream, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Liposomal Bupivacaine 266mg Knee Infiltration
  Liposomal Bupivacaine: administered via local tissue infiltration around the knee joint.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Liposomal Bupivacaine,: Liposomal Bupivacaine 266mg, Knee Infiltration
  Liposomal Bupivacaine: administered via local tissue infiltration around the knee joint.
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine, | Bupivacaine HCl | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.19 (7.59) | 62.29 (8.11) | 63.22 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 18 | 12 | 30
Region of Enrollment [Number; unit: Count of Participants]
  United States | 32 | 33 | 65
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 33.13 (4.53) | 32.57 (4.55) | 32.84 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity at Movement
Description: Pain intensity at maximum knee flexion measured using a 0-10 visual analog scale.
  Higher values represent a higher pain intensity or worse outcome.
Time Frame: 24hrs
Measure: Mean (95% Confidence Interval); unit: VAS Scale
Arm/Group | Liposomal Bupivacaine, | Bupivacaine HCl
Number analyzed (Participants) | 32 | 33
VAS Scale | 8.95 [8.42 to 9.48] | 7.91 [7.19 to 8.61]

2. Secondary Outcome: Pain Intensity at Rest
Description: as for outcome 1
Time Frame: 24hrs
Measure: Mean (95% Confidence Interval); unit: VAS Scale
Groups:
- Liposomal Bupivacaine: Liposomal Bupivacaine 266mg, Knee Infiltration
  Liposomal Bupivacaine: Administered via local tissue infiltration around the knee joint
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 32 | 33
VAS Scale | 5.08 [4.18 to 5.98] | 5.16 [4.17 to 6.14]

3. Secondary Outcome: Opioid Consumption
Time Frame: 24hrs
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 32 | 33
Morphine milligram equivalents | 28.91 [22.11 to 35.70] | 26.32 [20.60 to 32.03]

4. Secondary Outcome: Mean Plasma Bupivicaine Level
Time Frame: 72hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.04 (0.01) | 1.08 (0.40)

5. Secondary Outcome: Mean Plasma Bupivacaine Levels
Time Frame: 48hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposome Bupivacaine, | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.29 (0.19) | 1.76 (0.53)

6. Secondary Outcome: Mean Plasma Bupivacaine Level
Time Frame: 24hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.5 (0.16) | 1.16 (0.40)

7. Secondary Outcome: Mean Plasma Bupivacaine Level
Time Frame: 12hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.49 (0.23) | 0.74 (0.25)

8. Secondary Outcome: Mean Plasma Bupivacaine Level
Time Frame: 4hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.35 (0.18) | 0.44 (0.16)

9. Secondary Outcome: Mean Plasma Bupivacaine Level
Time Frame: 2hrs
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Standard Deviation); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.24 (0.1) | 0.29 (0.15)

10. Secondary Outcome: Mean Plasma Bupivacaine Level
Time Frame: Baseline
Population: Of the 32 and 33 participants in each arm 11 and 12 were allocated respectively to receive a blood draw
Measure: Mean (Full Range); unit: microgram per mL
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 11 | 12
microgram per mL | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 16/32 | 25/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=32) | Bupivacaine HCl (N=33)
PONV (Gastrointestinal disorders) | 7 | 10 — Postoperative nausea and vomiting
Hypotension (Nervous system disorders) | 1 | 8
Chest Pains (Cardiac disorders) | 0 | 1
Somnolence (General disorders) | 3 | 3
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 | 1
Knee Swelling (Injury, poisoning and procedural complications) | 2 | 1
headache (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No